CLINICAL TRIAL: NCT06564506
Title: Electroacupuncture for Preventing Postoperative Delirium in Older Adults Undergoing Total Knee Arthroplasty: a Multicentre Randomised Controlled Trial
Brief Title: Electroacupuncture for Preventing Postoperative Delirium in Older Adults Undergoing Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K2023-02-004/02
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Delirium
Keywords: Older adults; Electroacupuncture; Postoperative delirium; Total knee arthroplasty
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active electroacupuncture group (Experimental): Participants will receive 30 minutes of active electroacupuncture before anaesthesia induction. Experienced acupuncturists will administer electroacupuncture at Shenting (GV24, 0.5 cun [≈10 mm] above the anterior hairline midpoint) and bilateral Benshen (GB13, 3 cun [≈60 mm] lateral to GV24). After skin preparation and pad placement, patients will close their eyes. Needles will be inserted 20 to 24 mm into the subgaleal layer at a flat angle, then manually manipulated to elicit de qi sensations (eg, fullness, numbness and soreness). Electrodes attached to the needle handles will deliver stimulation for 30 minutes (2 Hz/15 Hz frequency, 1 mA intensity) to cause mild skin movement without pain.
  Interventions: Device: Disposable acupuncture needles (0.30 × 75 mm); Device: SDZ-V electroacupuncture devices
- Sham electroacupuncture group (Sham Comparator): Participants will receive 30 minutes of sham electroacupuncture before anaesthesia induction.The sham group will use non-acupuncture points: 20 mm above GV24 and 20 mm lateral to GB13. These points, in different dermatomes from true acupoints, minimise location-specific effects. The procedure will match the active group, excluding needle manipulation, de qi sensation and electrical output.
  Interventions: Device: Placebo needles (0.30 × 25 mm); Device: SDZ-V electroacupuncture devices

INTERVENTIONS:
Device: Disposable acupuncture needles (0.30 × 75 mm) — Disposable acupuncture needles (0.30 × 75 mm), placebo needles (0.30 × 25 mm) and SDZ-V electroacupuncture devices (Hwato, Suzhou Medical Supplies Factory Co Ltd, China) will be used. Electrodes attached to the needle handles will deliver stimulation for 30 minutes (2 Hz/15 Hz frequency, 1 mA intensity) to cause mild skin movement without pain.
  Arms: Active electroacupuncture group
Device: Placebo needles (0.30 × 25 mm) — Disposable acupuncture needles (0.30 × 75 mm), placebo needles (0.30 × 25 mm) and SDZ-V electroacupuncture devices (Hwato, Suzhou Medical Supplies Factory Co Ltd, China) will be used. Sham electroacupuncture will use blunt-tipped placebo needles without current output, which retract into their handles to simulate skin insertion.
  Arms: Sham electroacupuncture group
Device: SDZ-V electroacupuncture devices — Disposable acupuncture needles (0.30 × 75 mm), placebo needles (0.30 × 25 mm) and SDZ-V electroacupuncture devices (Hwato, Suzhou Medical Supplies Factory Co Ltd, China) will be used. Electrodes attached to the needle handles will deliver stimulation for 30 minutes (2 Hz/15 Hz frequency, 1 mA intensity) to cause mild skin movement without pain.

SUMMARY:
Electroacupuncture may improve cognitive function and altered consciousness, but its effect on postoperative delirium in older arthroplasty patients remains unexplored. This study aims to assess the efficacy of electroacupuncture in preventing postoperative delirium in older adults undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Electroacupuncture combines traditional acupuncture with electrical stimulation at specific body points. Recent clinical studies have shown promising results for acupuncture-related techniques in managing perioperative neurocognitive disorders. However, the efficacy of electroacupuncture in preventing postoperative delirium in elderly patients undergoing total knee arthroplasty remains unexplored.This randomised controlled trial aims to evaluate the efficacy of electroacupuncture in preventing postoperative delirium in elderly patients undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-90 years
* American Society of Anaesthesiologists (ASA) physical status class II or III
* Scheduled for elective unilateral total knee arthroplasty under general anesthesia

Exclusion Criteria:

* Baseline dementia or Mini-Mental State Examination (MMSE) score below 24
* Implanted electrical devices (eg, pacemakers, brain or spinal cord neurostimulator)
* Infection or abscess at any selected acupuncture point
* Severe hematopoietic or hemorrhagic disease
* Severe audio-visual impairments or inability to communicate in Mandarin
* Alcohol or illicit drug misuse disorder
* Current use of sedatives, antidepressants or glucocorticoids
* Received acupuncture or electroacupuncture within one month before surgery
* Any condition deemed unsafe or unsuitable by the research team

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1460 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium within the first three postoperative days | At least two hours postsurgery and twice daily (09:00-11:00 and 18:00-20:00) for three days
  The incidence of POD within the first three postoperative days will be assessed using the Confusion Assessment Method (CAM). The CAM evaluates four diagnostic features: (1) acute onset or fluctuating course, (2) inattention, (3) disorganised thinking and (4) altered consciousness. Delirium is diagnosed when features 1 and 2 are present, with either 3 or 4. Blinded investigators will assess for POD at least two hours postsurgery and twice daily (09:00-11:00 and 18:00-20:00) for three days.

SECONDARY OUTCOMES:
Delirium severity | At least two hours postsurgery and twice daily (09:00-11:00 and 18:00-20:00) for three days
  Delirium Rating Scale-Revised-98 (DRS-R-98); range 0-39, higher scores indicate greater severity
Delirium subtypes | At least two hours postsurgery and twice daily (09:00-11:00 and 18:00-20:00) for three days
  Richmond Agitation Sedation Scale (RASS); hypoactive (-3 to 0), hyperactive (+1 to +4) or mixed
Cognitive function | At 1, 3, 6 and 12 months postoperatively
  Abbreviated Mental Test Score (AMTS) via telephone at 1, 3, 6 and 12 months postoperatively
Anxiety and depression | Assessed preoperatively and daily for three days postoperatively
  Hospital Anxiety and Depression Scale (HADS); 14-item checklist (7 for anxiety, 7 for depression); each item scored 0-3; total score >8 suggests mild disorder, >10 moderate disorder
Postoperative pain | Assessed at 1, 3, 6, 12, 24, 36, 48, 60 and 72 hours postsurgery
  11-point Numerical Rating Scale (0 = no pain, 10 = worst pain imaginable) at rest and movement
Postoperative morphine consumption | During 72 hours postsurgery
  Cumulative morphine use and rescue analgesia recorded over 72 hours postsurgery
Recovery quality | Assessed daily for three days postoperatively
  Chinese version of the 15-item Quality of Recovery Questionnaire (QoR-15); range 0-150, higher scores indicate better recovery
Sleep quality | Assessed preoperatively and daily for three days postoperatively
  Richards-Campbell Sleep Questionnaire (RCSQ); higher mean scores indicate better sleep
Adverse events | through study completion, an average of 7 days
  Any adverse events during the study will be documented on the electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Yusheng Yao, MD, Principal Investigator — Fujian Provincial Hospital, China
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
The individual deidentified participant data, the study protocol, and the statistical analysis plan can be accessed from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 3 months after publication, until 5 years.